CLINICAL TRIAL: NCT01807767
Title: Prospective Evaluation of the Efficacy and Safety of Zortress (Everolimus)/Myfortic (Enteric Coated Mycophenolate Sodium) Conversion in High MELD Liver Transplantation
Brief Title: Myfortic in High MELD Liver Transplantation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: funding was withdrawn
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-0457; CRAD001HUS63T
Record Dates: First submitted 2013-03-06; First posted 2013-03-08 (Estimated); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: High Model for End-Stage Liver Disease (MELD) Score
MeSH Terms: interventions — Everolimus; Mycophenolic Acid; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Everolimus, Myfortic and Tacrolimus (Experimental): Tacrolimus discontinued (within 8 weeks of initiation of everolimus conversion).
  Everolimus 1mg BID started (targeted trough 6-12ng/mL). Patients must have an everolimus concentration between 6-12ng/mL before tacrolimus is discontinued.
  Myfortic 360-720 mg BID
  Interventions: Drug: Everolimus, Myfortic and Tacrolimus
- Myfortic and Tacrolimus (Other): Normal Care: Myfortic BID 360-720 mg Tacrolimus (5-12ng/mL)
  Interventions: Drug: Myfortic and Tacrolimus

INTERVENTIONS:
Drug: Everolimus, Myfortic and Tacrolimus — Tacrolimus discontinued (within 8 weeks of initiation of everolimus conversion).
  Everolimus 1mg BID started (targeted trough 6-12ng/mL). Patients must have an everolimus concentration between 6-12ng/mL before tacrolimus is discontinued.
  Myfortic 360-720 mg BID
  Other Names: Everolimus: Zortress, Certican, Afinitor; Myfortic: CellCept; Tacrolimus: FK-506, fujimycin, Prograf, Advagraf, Protopic
  Arms: Everolimus, Myfortic and Tacrolimus
Drug: Myfortic and Tacrolimus — Myfortic BID 360-720 mg Tacrolimus (5-12ng/mL)
  Other Names: Myfortic: CellCept; Tacrolimus: FK-506, fujimycin, Prograf, Advagraf, Protopic
  Arms: Myfortic and Tacrolimus

SUMMARY:
The objective of the study is to determine the efficacy and safety of Everolimus conversion in liver transplantation. Most large US liver centers transplant patients with high Model for End-Stage Liver Disease (MELD) scores. However, many of the sponsored liver transplant trials in the US do not include patients with high MELD scores making it difficult to extrapolate these trial data to the patients cared for at larger liver transplant centers. The greatest potential benefit of mammalian target of rapamycin (mTOR) inhibitors is the avoidance of the side-effects of calcineurin-inhibitors, namely, renal insufficiency, diabetes and hypertension. Therefore, this protocol is designed to study the efficacy and safety of everolimus and Myfortic in liver transplant patients with high MELD scores at two large centers with a vast experience in the administration of mTOR inhibitors.

ELIGIBILITY:
Inclusion Criteria:

Patients must give written informed consent before any assessment is performed.

1. MELD ≥ 25.
2. Recipients who are 18-70 years of age of a primary or secondary liver transplant from a deceased donor.
3. Allograft is functioning at an acceptable level by the time of randomization as defined by the Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), Total Bilirubin levels ≤3 times Upper Limit of Normal (ULN), and Alkaline Phosphatase (AlkP) levels ≤ 5 times ULN.
4. Ability and willingness to provide written informed consent and adhere to study regimen.
5. Patients who are able to take oral medication at time of randomization. Glomerular Filtration Rate (GFR) ≥ 30 ml/min.

Exclusion Criteria:

1. Patients receiving 3rd transplants
2. Fulminant hepatic failure
3. Living donor transplants
4. Donation after Cardiac Death (DCD) donors or split grafts
5. Active infection or hemodynamic instability at the time of transplant
6. Renal replacement therapy for clearance within 7 days prior to randomization
7. Presence of thrombosis via Doppler ultrasound of the major hepatic arteries, major hepatic veins, portal vein and inferior vena cava.
8. An episode of acute rejection that required antibody therapy or more than one steroid sensitive episode of acute rejection prior to randomization. This includes patients who have not completed steroid treatment for acute rejection within 7 days prior to randomization.
9. Spot urine protein/creatinine ratio > 1g/24h at time of randomization
10. Combined liver/kidney transplant
11. Patients who have severe hypercholesterolemia (>350 mg/dL) or Patients with platelet count < 50,000 at time of randomization
12. Patients with an Absolute neutrophil count (ANC) of < 1,000 or White Blood Count (WBC) of <2,000 at time of randomization
13. Patients with hemoglobin <6g/dL
14. Patients who are unable to take oral medication at time of randomization
15. Patients with clinically significant systemic infection requiring active use of IV antibiotics, anti-virals, or anti-fungals
16. Patients who are in a critical care setting at the time of randomization requiring life support measures such as mechanical ventilation, dialysis, requirement of vasopressor agents
17. Known intolerance to tacrolimus or everolimus or Myfortic.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-03; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
proven acute rejection | 12 months
  1. To evaluate the use of a calcineurin-free immunosuppressive regimen utilizing concentration-controlled everolimus and mycophenolic acid (Myfortic) (Arm #12), in order to compare rates of the composite efficacy endpoint (biopsy proven-acute rejection, graft loss, and death) to the rates in the CNI-containing control arm (Arm #21) at 12 months post conversion to everolimus.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Zimmerman, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States